CLINICAL TRIAL: NCT06981741
Title: Phase I/IIa Study to Test the Safety and Efficacy of MSC From Umbilical Cord Tissue (UC-MSC) for the Treatment of Cartilage Damage in the Knee Joint
Brief Title: Safety and Efficacy of hUC-MSC for the Treatment of Cartilage Damage in the Knee Joint
Acronym: BPCC001
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BIONCaRT GmbH (Industry)
Collaborators: KKS Netzwerk (Network); Fraunhofer Institute for Cell Therapy and Immunology IZI (Unknown); Polski Bank Komorek Macierzystych JSC (PBKM) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MesemCart2Clinic - BP CC 001; 2024-517684-23-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Cartilage Damage
Keywords: knee; cartilage; mesenchymal stromal cells; mesenchymal stem cells; UC-MSC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational Product Arm (Experimental): Participants in this arm will undergo arthroscopic or minimally invasive knee surgery, during which the investigational product - mesenchymal stromal cells (MSCs) derived from umbilical cord tissue (MesemCart) - will be applied once directly to the cartilage defect. All patients will receive the same treatment and will be monitored for safety and initial efficacy outcomes over a period of 24 months.
  Interventions: Biological: BP CC 001

INTERVENTIONS:
Biological: BP CC 001 — 10-20 x 10^6 UC-MSC in 1 ml suspension, applied to a collagen carrier structure (Chondro-Gide®)

SUMMARY:
Testing the safety and efficacy of MSC from umbilical cord tissue (UC-MSC) for the treatment of cartilage damage in the knee joint

DETAILED DESCRIPTION:
All patients who provide written informed consent after receiving detailed information about the study and its potential risks will undergo a screening to assess eligibility. This is a prospective, multicenter, single-arm, open-label clinical trial. On Visit 1 (Day 0), eligible patients will receive knee surgery with a one-time application of the investigational product to the cartilage defect. Follow-up visits over a two-year period will be conducted at regular intervals to monitor the safety of the investigational product and to collect initial data on its efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any gender with an age from ≥ 18 years to ≤ 60 years
* Clinical indication for a surgical cartilage regeneration procedure
* Symptomatic grade III/IV cartilage defect according to ICRS or osteochondral defect with a maximum depth of 3 mm
* A cartilage defect requiring treatment with a defect size of 2-6 cm² on the femoral condyles or patella or trochlea
* Affected and contralateral knee (if known): Kellgren-Lawrence (K/L) osteoarthritis severity < grade III
* KOOS pain sub-score of ≤ 70 (out of max. 100) in the affected knee joint and > 80 (out of max. 100) in the contralateral knee joint measured without taking analgesics within the last 24 hours
* BMI < 35 kg/m²
* Written informed consent of the participant, also regarding alternative procedures such as cartilage transplantation (MACT) or matrix-augmented bone marrow stimulation (BMS, AMIC)

Exclusion Criteria:

* Clinical indication explicitly for a cartilage regeneration procedure other than the intended study treatment
* Known varus or valgus malalignment of the affected leg of ≥ 5°
* Antero-posterior or medio-lateral instability
* Meniscus loss of more than 20% in the affected compartment
* Patella instability
* Simultaneous surgery on other joint structures (cruciate ligament replacement, meniscus suture, partial meniscus resection > 20%, osteotomy)
* Simultaneous higher-grade (ICRS grade III/IV) cartilage damage on the corresponding joint surfaces to the treated cartilage damage ("kissing lesions")
* Osteoarthritis Kellgren-Lawrence (K/L) grade III or IV
* Arthrofibrosis
* Metabolic arthropathy
* Collagenosis
* Autoimmune disease
* Tumor disease within the last 5 years
* Neuromuscular disease
* Peripheral arterial occlusive disease
* Intra-articular application of hyaluronic acid or glucocorticoids or platelet concentrates within the last 6 months
* Joint replacement in the contra-lateral knee or hip within the last 12 months
* Rheumatoid arthritis or other inflammatory diseases such as autoimmune diseases, seronegative spondyloarthritis, gout, pseudogout
* Previous fracture in the affected knee joint
* Osteoporosis
* Contraindications against the planned operation under general anesthesia
* Relevant secondary diseases that increase the risk of surgery, e.g. cardiac insufficiency, coronary heart disease, coagulation disorders, diabetes mellitus, liver cirrhosis, renal insufficiency, etc.
* History of known hypersensitivity to porcine collagens, human albumin, glucose or components of fibrin adhesives used in orthopaedics or surgery
* Simultaneous participation in another interventional clinical trial (incl. within the last 4 weeks prior to inclusion)
* Addiction or other illnesses that do not allow the person concerned to assess the nature, scope and possible consequences of the clinical trial (lack of capacity to consent)
* Indications that the patient is unlikely to adhere to the protocol (e.g. lack of compliance)
* Persons who are placed in an institution by court or official order
* Persons who are dependent on the sponsor
* Pregnant or breastfeeding women
* Women of childbearing age, except women who meet the following criteria:

  1. Post-menopausal (12 months natural amenorrhea)
  2. Post-operative (6 weeks after bilateral ovariectomy with or without hysterectomy or bilateral salpingectomy)
  3. Presence of a negative pregnancy test (urine, not older than 14 days on the day of surgery) and willingness to regularly and correctly use a contraceptive method with a Pearl Index < 1 % per year:

     3.1 Combined (oestrogen and progestogen-containing) hormonal contraception 3.2 Hormonal contraception containing progestogens (oral, injected, implanted) 3.3 IUD (hormonal IUD, copper IUD)
  4. Sexual abstinence
  5. Vasectomy of the partner

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a serious adverse event within 24 months after surgery | within 24 months after surgery

SECONDARY OUTCOMES:
Regeneration of damaged cartilage measured using the MOCART score | 12 months after surgery
  The MOCART (Magnetic Resonance Observation of Cartilage Repair Tissue) scoring system ranges from 0 to 100. A score of 0 indicates no repair, while 100 represents an excellent cartilage defect repair.
Relative change in pain in the knee joint compared to the initial value before the operation measured using the KOOS Pain Subscore | 12 and 24 months after the operation
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) ranges from 0 to 100, where 0 represents extreme knee problems and 100 represents no knee problems.
Relative change in knee-related quality of life compared to pre-surgery baseline measured by KOOS-QoL subscore | 12 and 24 months after surgery
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) ranges from 0 to 100, where 0 represents extreme knee problems and 100 represents no knee problems.
Relative change in symptoms and stiffness compared to pre-surgery baseline as measured by KOOS symptom subscore | 12 and 24 months after surgery
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) ranges from 0 to 100, where 0 represents extreme knee problems and 100 represents no knee problems.
Relative change in activities of daily living compared to pre-surgery baseline measured by KOOS-ADL subscore | 12 and 24 months after surgery
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) ranges from 0 to 100, where 0 represents extreme knee problems and 100 represents no knee problems.
Relative change in physical resilience during sporting activities after the operation compared to the initial value before the operation measured using the KOOS-Sport/Rec-Subscore | 12 and 24 months
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) ranges from 0 to 100, where 0 represents extreme knee problems and 100 represents no knee problems.
Description of all adverse events (AE, AR, SAE, SAR, SUSAR) with regard to severity (assessed according to NCI-CTCAE V 5.0), causality, outcome | within 24 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Lützner, Prof.Dr.med., Principal Investigator — UniversitätsCentrum für Orthopädie, Unfall- & Plastische Chirurgie, Universitätsklinikum Carl Gustav Carus, TU Dresden
Locations (7):
- Germany (7):
  - Klinikum Altenburger Land, Klinik für Orthopädie und Unfallchirurgie, Altenburg
  - St. Nikolaus Stifts-Hospital, Andernach
  - Sozialstiftung Bamberg Klinikum am Bruderwald, Klinik für Orthopädie und Unfallchirurgie, Bamberg
  - Evangelisches Waldkrankenhaus Spandau, Berlin
  - GFO Kliniken Niederrhein, St. Vinzenz Hospital Dinslaken, Dinslaken
  - UniversitätsCentrum für Orthopädie, Unfall- & Plastische Chirurgie, Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Maria-Josef-Hospital Greven, Klinik für Unfallchirurgie und Orthopädie, Greven

IPD SHARING:
Plan to Share IPD: Undecided